CLINICAL TRIAL: NCT06650449
Title: APP: Modelo De Intervención En Salud Mental En Personal Sanitario
Brief Title: APP: Mental Health Intervention Model for Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labora (Other)
Responsible Party: Principal Investigator, Marco Antonio Faytong Haro, Research Professor, Universidad de Especialidades Espiritu Santo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LIDE-2022-001
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorders; Anxiety Disorders; Mental Health
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study follows a case-control interventional model. Participants are divided into two groups: an intervention group using a mobile app based on Cognitive Behavioral Therapy (CBT) techniques, and a control group receiving no intervention. The app delivers weekly tasks over a 3-month period aimed at reducing emotional distress and depressive symptoms in healthcare workers. Both groups will be assessed at the start and end of the study using the PHQ-9 and GHQ-12 questionnaires to evaluate changes in mental health. The design allows for a comparison of mental health outcomes between those who receive the app-based intervention and those who do not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Mobile App-Based Mental Health Support) (Experimental): Participants in this group will use a mobile app designed to deliver cognitive-behavioral therapy (CBT) techniques over a 3-month period. The app provides 12 weekly tasks aimed at reducing emotional distress and depressive symptoms. Tasks include exercises on emotional regulation, coping strategies, and mindfulness. Progress is tracked via the app, and participants will complete the PHQ-9 and GHQ-12 questionnaires at the start and end of the intervention.
  Interventions: Other: Mobile App-Based Mental Health Support
- Control Group (No Intervention) (No Intervention): Participants in this group will not receive any mental health intervention during the study period. They will complete the PHQ-9 and GHQ-12 questionnaires at the start and end of the 3-month period to assess changes in emotional distress and depressive symptoms for comparison with the intervention group.

INTERVENTIONS:
Other: Mobile App-Based Mental Health Support — This intervention uses a mobile application designed to deliver Cognitive Behavioral Therapy (CBT) techniques. The app provides 12 weekly tasks aimed at reducing emotional distress and depressive symptoms in healthcare workers. Tasks include exercises on emotional regulation, coping strategies, and mindfulness. Participants receive notifications to encourage task completion, and the app tracks progress over the 3-month period. At the start and end of the study, participants will complete the PHQ-9 and GHQ-12 questionnaires to assess their mental health status.
  Arms: Intervention Group (Mobile App-Based Mental Health Support)

SUMMARY:
This study, titled "APP: Mental Health Intervention Model for Healthcare Workers," aims to evaluate the effectiveness of a mobile app-based intervention to reduce emotional distress and symptoms of depression among healthcare workers at Hospital León Becerra in Milagro, Ecuador. The app, designed with cognitive-behavioral techniques, offers weekly tasks to improve mental health over a three-month period. The study follows a case-control design, with initial and follow-up evaluations using the PHQ-9 and GHQ-12 questionnaires to assess mental health status. The expected outcome is a significant reduction in emotional distress and depression symptoms among the participants.

DETAILED DESCRIPTION:
Detailed Description:

This study, titled "APP: Mental Health Intervention Model for Healthcare Workers," seeks to evaluate a novel mobile app-based intervention aimed at addressing mental health challenges among healthcare professionals at Hospital León Becerra in Milagro, Ecuador. The intervention leverages Cognitive Behavioral Therapy (CBT) techniques to mitigate emotional distress and reduce symptoms of depression. This approach offers a scalable, flexible, and low-cost solution to support mental well-being in healthcare environments, particularly in response to the increased psychological strain caused by the COVID-19 pandemic.

Study Rationale and Theoretical Framework:

Healthcare workers are often exposed to stressors that lead to cumulative mental health burdens, including extended working hours, emotional labor, and the pressure of making life-or-death decisions in real time. The added impact of the pandemic has exacerbated these stressors, leading to a rise in reported cases of burnout, anxiety, and depression. In resource-limited settings, where access to mental health services is often restricted due to logistical, financial, or cultural barriers, mobile health (mHealth) interventions offer a promising solution.

The intervention model of this study is grounded in Cognitive Behavioral Therapy (CBT), a well-established psychotherapeutic approach with a strong evidence base for treating depression and anxiety. CBT works by helping individuals identify and challenge negative thought patterns, develop emotional regulation techniques, and engage in behaviors that improve mood and well-being. In digital form, CBT maintains its efficacy and can be delivered asynchronously, making it ideal for busy healthcare workers who need flexibility in how and when they access mental health support.

Intervention Model and App Features:

The mobile app used in this study has been specifically designed to incorporate core components of CBT, including cognitive restructuring, behavioral activation, and emotional regulation strategies. It delivers 12 weekly tasks that participants are expected to complete over a three-month period. The app has been developed with healthcare professionals in mind, considering the high-demand nature of their work and their need for accessible, short, and impactful mental health tools.

Each weekly task focuses on a different aspect of CBT and is structured to promote cognitive reframing, emotional awareness, and behavior change. Examples of tasks include:

Week 1-3: Introducing participants to the basics of CBT and guiding them in identifying negative thought patterns that contribute to emotional distress.

Week 4-6: Implementing emotional regulation strategies, teaching participants how to manage stress, anxiety, and sadness through mindfulness and relaxation techniques.

Week 7-9: Engaging in behavioral activation, encouraging participants to take actionable steps to improve their mood, such as goal setting and increasing engagement in pleasurable activities.

Week 10-12: Reinforcing coping strategies and relapse prevention techniques to help participants maintain their mental well-being after completing the program.

The app features include:

Interactive Tasks: Participants complete guided exercises within the app that allow them to apply CBT techniques to their own experiences.

Reminders and Prompts: Automated notifications remind participants to complete their weekly tasks, improving adherence to the intervention.

Progress Tracking: Participants can track their progress over time, reviewing completed tasks and assessing improvements in their emotional state.

Resource Library: The app provides access to educational materials on stress management, self-care, and coping mechanisms that healthcare workers can access at their convenience.

Study Design:

The case-control study design allows for a robust evaluation of the app's effectiveness. Participants are randomized into either the intervention group, which will use the app, or the control group, which will not receive the app intervention during the study period. This design allows for clear comparison between groups, controlling for natural fluctuations in mental health that might occur over time without the intervention.

The primary objective is to assess the effectiveness of the app in reducing symptoms of depression (as measured by the PHQ-9) and emotional distress (as measured by the GHQ-12). The secondary objectives include evaluating user engagement with the app, user satisfaction, and the feasibility of scaling the intervention to other healthcare settings.

Implementation and Technology Integration:

The mobile app will be implemented in a user-friendly manner, compatible with both Android and iOS devices. Participants will be provided with a secure download link, and the app will include a brief tutorial to help users familiarize themselves with its features. Data collected through the app (including questionnaire responses and engagement metrics) will be encrypted and securely transmitted to a central server for analysis, ensuring participant confidentiality and compliance with data privacy regulations.

To facilitate high engagement, the app has been designed with busy healthcare professionals in mind, offering flexibility in when and where they complete their weekly tasks. The app's design also includes built-in mechanisms to identify users who may need more intensive mental health support. For example, if a participant reports severely elevated depression scores during any task, the app will trigger an alert, prompting the research team to reach out and offer additional support or referrals to mental health services.

Data Collection and Analysis Plan:

The primary data for this study will be collected through the PHQ-9 and GHQ-12 questionnaires, administered at baseline (T0) and three months post-intervention (T1). These tools are internationally recognized and validated for assessing depression and emotional distress, respectively. In addition to self-reported mental health outcomes, user engagement data (such as task completion rates and time spent on the app) will be automatically tracked by the app.

Data will be analyzed using both descriptive and inferential statistics:

Descriptive statistics will summarize baseline characteristics of the participants, including age, gender, professional role, and prior mental health diagnoses.

Independent t-tests will be used to compare the mean change in PHQ-9 and GHQ-12 scores between the intervention and control groups.

Multivariate logistic regression models will be employed to adjust for potential confounders, such as age, profession, education level, and prior mental health status. These models will help isolate the effect of the intervention from other factors that may influence mental health outcomes.

User engagement metrics will be analyzed to determine adherence to the intervention and its correlation with changes in mental health outcomes. This will involve examining the relationship between app usage (e.g., number of completed tasks) and reductions in PHQ-9 and GHQ-12 scores.

Ethical Considerations and Feasibility:

The study protocol has been reviewed and approved by the ethics committee at Hospital León Becerra, and informed consent will be obtained from all participants before their enrollment. Participants will be fully informed about the study's objectives, their right to withdraw at any point, and the confidentiality measures in place. Mental health support will be available to participants who exhibit elevated levels of distress during the study, ensuring their well-being is prioritized.

This study represents a critical step in assessing the feasibility and effectiveness of mHealth interventions in healthcare settings. The findings will not only contribute to the understanding of digital mental health tools but also provide practical insights into how these tools can be integrated into the daily lives of healthcare professionals, helping to mitigate the mental health crisis facing this population.

ELIGIBILITY:
Inclusion Criteria:

Must be a healthcare worker (doctor, nurse, therapist, etc.) employed at Hospital León Becerra in Milagro, Ecuador.

Must have been working at the hospital for at least 12 months. Aged 18 years or older. Willing to participate in the study and able to provide informed consent.

Exclusion Criteria:

Healthcare workers on leave, incapacity, or vacation during the study period. Those who do not wish to participate in the study. Individuals who no longer work at Hospital León Becerra.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire) | 3 months (at baseline and after completion of the 12-week intervention).
  The PHQ-9 (Patient Health Questionnaire-9) is a widely used, brief self-administered tool for screening, diagnosing, monitoring, and measuring the severity of depression. It is based on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM) and includes nine items that reflect the core symptoms of depression.
  Each of the nine items corresponds to a symptom of depression, and respondents are asked to rate how often they have been bothered by each symptom over the past two weeks. The response options are:
  0: Not at all
  1. Several days
  2. More than half the days
  3. Nearly every day The total score ranges from 0 to 27, with higher scores indicating more severe depression.
GHQ-12 (General Health Questionnaire) | 3 months (at baseline and after completion of the 12-week intervention).
  GHQ-12 (General Health Questionnaire-12) with Likert Scoring The GHQ-12 with Likert scoring is designed to assess the level of psychological distress by assigning a numerical value to each response on a 4-point scale. This method allows for more nuanced analysis of the severity of mental health issues, rather than just categorizing them as "present" or "absent" as in the bimodal scoring method.
  Likert Scoring Scale:
  For each of the 12 items, responses are scored as follows:
  0: Not at all
  1. No more than usual
  2. Rather more than usual
  3. Much more than usual This creates a continuous scale where the total score can range from 0 to 36, with higher scores indicating more severe distress.
  Example Items and Scoring:
  Have you recently been able to concentrate on whatever you're doing?
  Not at all (0) No more than usual (1) Rather more than usual (2) Much more than usual (3) Have you recently lost much sleep over worry?
  Not at all (0) No more than usual (1) Rather more than usual (2) Mu

CONTACTS AND LOCATIONS:
Locations (1):
- UEES, Samborondón, Ecuador

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns regarding confidentiality and privacy of healthcare workers' sensitive mental health information. The study data will be securely stored, and only aggregated results will be published, ensuring that participants' identities remain confidential. Sharing individual data could pose a risk of identifying participants, especially in a specific healthcare setting.